CLINICAL TRIAL: NCT04194021
Title: Demographic, Clinical, and Laboratory Characteristics and Outcomes of Patients Who Ever Received Etravirine and/or Darunavir - Multi-country Data Abstraction
Brief Title: Characteristics and Outcomes of Patients Who Received Etravirine and/or Darunavir
Acronym: NewHorizon
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: EG0205
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Antiretroviral therapy; Darunavir; Etravirine; Treatment-experienced HIV; Pediatrics; Adolescents; Young people; Drug resistance mutations; Cameroon; Eswatini; Ethiopia; Kenya; Lesotho; Nigeria; Uganda; Zambia; Zimbabwe; Viral load; Protease inhibitor; Non-nucleoside reverse transcriptase inhibitor
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The objectives of this data collection activity are to:

1. Describe the baseline demographics, clinical and laboratory profile of patients who ever received darunavir (DRV) and/or etravirine (ETR), at the time of initiation on DRV and/or ETR;
2. Describe the clinical and laboratory profile of patients who ever received DRV and/or ETR every 6 months from the first data collection point through 2021;
3. Describe dynamics in HIV drug resistance mutations among patients who fail treatment on new regimens including DRV and/or ETR;
4. Describe demographics, clinical and laboratory profile of young adults who transition out of the donation program after the age of 25 years at 12 months after their transition.

DETAILED DESCRIPTION:
Janssen, the Elizabeth Glaser Pediatric AIDS Foundation (EGPAF), the Partnership for Supply Chain Management (PFSCM), the Collaborative Initiative for Pediatric HIV Education and Research (CIPHER) of the International AIDS Society (IAS), and Right to Care have partnered to implement the New Horizons Collaborative to improve and scale-up pediatric HIV/AIDS care and treatment through increased awareness, research, health systems strengthening, and improved access to HIV/AIDS medicines. A primary source of darunavir (DRV) and etravirine (ETR) for pediatric populations in sub-Saharan Africa is through the New Horizons DRV/ETR Donation Program, which was launched in 2014. Under this program, Janssen provides DRV and/or ETR free of charge to eligible national HIV/AIDS programs in sub-Saharan Africa, for use in children and adolescents up to 25 years of age.

Countries currently participating in the New Horizons Collaborative include: Cameroon, Eswatini, Ethiopia, Kenya, Lesotho, Nigeria, Rwanda, Uganda, Zambia, and Zimbabwe. Any country that applies and is approved for receipt of donated product will become eligible for this study when they begin offering donated product to patients.

Prior to the inception of the New Horizons Collaborative, no multi-country data were collected regarding the demographic or clinical characteristics of the target patient population (i.e., children, adolescents, and young people < 25 years in need of second- or third-line HIV/AIDS treatment). Therefore, the current activity proposes to collect cross-sectional demographic and clinical data at baseline and every six months for patients receiving DRV and/or ETR across participating New Horizons countries. This activity will comprise data abstraction of key demographic, clinical, laboratory and case history indicators and outcomes on each patient who ever received DRV and/or ETR.

ELIGIBILITY:
Inclusion Criteria:

* Ever received darunavir and/or etravirine.
* Under age 25.
* Residing in any of the following countries: Cameroon, Ethiopia, Eswatini, Kenya, Lesotho, Nigeria, Rwanda, Uganda, Zambia, and Zimbabwe.

Exclusion Criteria:

* Above age 25.
* Residing in a country not participating in the New Horizons Collaborative.

Max Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients who ever received darunavir and/or etravirine before turning age 25 and residing in the following countries: Cameroon, Eswatini, Kenya, Lesotho, Nigeria, Rwanda, Uganda, Zambia, Zimbabwe.
Sampling Method: Non-Probability Sample
Enrollment: 871 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical profile of patients who ever received darunavir and/or etravirine | At initiation of darunavir and/or etravirine, thereafter every six months to the end of 2021, 12 months after turning age 25
  Clinical and laboratory profiles of patients who ever received darunavir and/or etravirine

SECONDARY OUTCOMES:
Demographic profile of patients who ever received darunavir and/or etravirine | At initiation of darunavir and/or etravirine
  Age and gender of patients who ever received darunavir and/or etravirine
Dynamics in HIV drug resistance mutations | At initiation of darunavir and/or etravirine, thereafter every six months to the end of 2021, 12 months after turning age 25
  Dynamics in HIV drug resistance mutations among patients who fail treatment

CONTACTS AND LOCATIONS:
Overall Officials: Appolinaire Tiam, MBChB, MMed, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (5):
- Elizabeth Glaser Pediatric AIDS Foundation/Cameroon, Yaoundé, Centre Region, Cameroon
- Elizabeth Glaser Pediatric AIDS Foundation/Eswatini, Mbabane, Hhohho Region, Eswatini
- Elizabeth Glaser Pediatric AIDS Foundation/Kenya, Nairobi, Kenya
- Elizabeth Glaser Pediatric AIDS Foundation/Lesotho, Maseru, Lesotho
- Elizabeth Glaser Pediatric AIDS Foundation/Uganda, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clavel F, Hance AJ. HIV drug resistance. N Engl J Med. 2004 Mar 4;350(10):1023-35. doi: 10.1056/NEJMra025195. No abstract available. PMID 14999114
- [Background] Petersen ML, van der Laan MJ, Napravnik S, Eron JJ, Moore RD, Deeks SG. Long-term consequences of the delay between virologic failure of highly active antiretroviral therapy and regimen modification. AIDS. 2008 Oct 18;22(16):2097-106. doi: 10.1097/QAD.0b013e32830f97e2. PMID 18832873
- [Background] Vaz P, Augusto O, Bila D, Macassa E, Vubil A, Jani IV, Pillon R, Sandstrom P, Sutherland D, Giaquinto C, Jordan MR, Bertagnolio S. Surveillance of HIV drug resistance in children receiving antiretroviral therapy: a pilot study of the World Health Organization's generic protocol in Maputo, Mozambique. Clin Infect Dis. 2012 May;54 Suppl 4(Suppl 4):S369-74. doi: 10.1093/cid/cis006. PMID 22544205
- [Background] Puthanakit T, Aurpibul L, Oberdorfer P, Akarathum N, Kanjanavanit S, Wannarit P, Sirisanthana T, Sirisanthana V. Sustained immunologic and virologic efficacy after four years of highly active antiretroviral therapy in human immunodeficiency virus infected children in Thailand. Pediatr Infect Dis J. 2007 Oct;26(10):953-6. doi: 10.1097/INF.0b013e318125720a. PMID 17901804
- [Background] Bolton-Moore C, Mubiana-Mbewe M, Cantrell RA, Chintu N, Stringer EM, Chi BH, Sinkala M, Kankasa C, Wilson CM, Wilfert CM, Mwango A, Levy J, Abrams EJ, Bulterys M, Stringer JS. Clinical outcomes and CD4 cell response in children receiving antiretroviral therapy at primary health care facilities in Zambia. JAMA. 2007 Oct 24;298(16):1888-99. doi: 10.1001/jama.298.16.1888. PMID 17954540
- [Background] Sutcliffe CG, van Dijk JH, Bolton C, Persaud D, Moss WJ. Effectiveness of antiretroviral therapy among HIV-infected children in sub-Saharan Africa. Lancet Infect Dis. 2008 Aug;8(8):477-89. doi: 10.1016/S1473-3099(08)70180-4. PMID 18652994
- [Background] Reddi A, Leeper SC, Grobler AC, Geddes R, France KH, Dorse GL, Vlok WJ, Mntambo M, Thomas M, Nixon K, Holst HL, Karim QA, Rollins NC, Coovadia HM, Giddy J. Preliminary outcomes of a paediatric highly active antiretroviral therapy cohort from KwaZulu-Natal, South Africa. BMC Pediatr. 2007 Mar 17;7:13. doi: 10.1186/1471-2431-7-13. PMID 17367540
- [Background] Katabira ET, Oelrichs RB. Scaling up antiretroviral treatment in resource-limited settings: successes and challenges. AIDS. 2007 Jul;21 Suppl 4:S5-10. doi: 10.1097/01.aids.0000279701.93932.ef. No abstract available. PMID 17620753
- [Background] Janssens B, Raleigh B, Soeung S, Akao K, Te V, Gupta J, Vun MC, Ford N, Nouhin J, Nerrienet E. Effectiveness of highly active antiretroviral therapy in HIV-positive children: evaluation at 12 months in a routine program in Cambodia. Pediatrics. 2007 Nov;120(5):e1134-40. doi: 10.1542/peds.2006-3503. Epub 2007 Oct 22. PMID 17954553
- [Background] Arasteh K, Yeni P, Pozniak A, Grinsztejn B, Jayaweera D, Roberts A, Hoy J, De Meyer S, Vangeneugden T, Tomaka F. Efficacy and safety of darunavir/ritonavir in treatment-experienced HIV type-1 patients in the POWER 1, 2 and 3 trials at week 96. Antivir Ther. 2009;14(6):859-64. doi: 10.3851/IMP1301. PMID 19812449
- [Background] Katlama C, Clotet B, Mills A, Trottier B, Molina JM, Grinsztejn B, Towner W, Haubrich R, Nijs S, Vingerhoets J, Woodfall B, Witek J. Efficacy and safety of etravirine at week 96 in treatment-experienced HIV type-1-infected patients in the DUET-1 and DUET-2 trials. Antivir Ther. 2010;15(7):1045-52. doi: 10.3851/IMP1662. PMID 21041921
- [Background] Imaz A, Llibre JM, Mora M, Mateo G, Camacho A, Blanco JR, Curran A, Santos JR, Caballero E, Bravo I, Gaya F, Domingo P, Rivero A, Falco V, Clotet B, Ribera E. Efficacy and safety of nucleoside reverse transcriptase inhibitor-sparing salvage therapy for multidrug-resistant HIV-1 infection based on new-class and new-generation antiretrovirals. J Antimicrob Chemother. 2011 Feb;66(2):358-62. doi: 10.1093/jac/dkq432. Epub 2010 Dec 14. PMID 21172789
- [Background] Fagard C, Colin C, Charpentier C, Rami A, Jacomet C, Yeni P, Vittecoq D, Katlama C, Molina JM, Descamps D, Chene G, Yazdanpanah Y; ANRS 139 TRIO Trial Group. Long-term efficacy and safety of raltegravir, etravirine, and darunavir/ritonavir in treatment-experienced patients: week 96 results from the ANRS 139 TRIO trial. J Acquir Immune Defic Syndr. 2012 Apr 15;59(5):489-93. doi: 10.1097/QAI.0b013e31824bb720. PMID 22293546
- [Background] Corrigan B, Mukui I, Mulenga L, Mthethwa N, Letsie M, Bruno S, Rakhmanina N. Characteristics of Treatment-experienced HIV-infected African Children and Adolescents Initiating Darunavir and/or Etravirine-based Antiretroviral Treatment. Pediatr Infect Dis J. 2018 Jul;37(7):669-672. doi: 10.1097/INF.0000000000001843. PMID 29140932

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT04194021/Prot_SAP_000.pdf